CLINICAL TRIAL: NCT01794234
Title: Efficacy and Safety of Peginterferon Alfa-2a (40 KD) in Chronic Hepatitis B Patients, Who Have Failed Anti-viral Treatment With Nucleoside (Nucleotide) Analogues - an Observational Study in Real-life Clinical Practice
Brief Title: An Observational Study of Pegasys (Peginterferon Alfa-2a) in Patients With Chronic Hepatitis B Who Have Failed Antiviral Treatment With Nucleoside (Nucleotide) Analogues
Status: Terminated | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28346
Record Dates: First submitted 2013-02-15; First posted 2013-02-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the efficacy and safety of Pegasys (peginterferon alfa-2a) in patients with chronic hepatitis B who have failed antiviral treatment with nucleoside (nucleotide) analogues. Data will be collected from patients treated according to the current Summary of Product Characteristics and local standard of care and regulations during 48 weeks of treatment and 24 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Positive HBsAg for more than 6 months before assignment to treatment with Pegasys
* Detectable HBV DNA (as measured by PCR)
* HBeAg positive and negative patients
* Patients previously treated with nucleoside (nucleotide) analogues who have failed antiviral treatment and have been assigned to treatment with Pegasys according to the local therapeutic standard
* Elevated serum alanine aminotransferase (ALT)
* Chronic hepatitis B confirmed by liver biopsy or non-invasive assessment (FibroScan), ARFI, FibroTest) or by clinical evaluation

Exclusion Criteria:

* Contraindications to treatment with Pegasys according to the Summary of Product Characteristics
* Hepatocellular carcinoma and/or severe hepatic dysfunction or decompensated cirrhosis of the liver
* Immunosuppression, immunomodulatory or chemotherapy within the last 6 months prior to start of Pegasys treatment
* Planned other than Pegasys antiviral treatment during Pegasys therapy
* Chronic liver disease other than chronic hepatitis B
* Pregnant or breast-feeding women
* Inadequate hematologic function
* Autoimmunology disorders
* Co-infection with chronic hepatitis C or HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B initiated on therapy with Pegasys
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Efficacy: HBsAg seroclearance/seroconversion rate at the end of Week 72 (48 weeks of treatment and 24 weeks of follow-up) | approximately 2.5 years

SECONDARY OUTCOMES:
HBs levels in correlation with treatment outcome | approximately 2.5 years
For HBeAg positive patients: Proportion of patients with HBeAg loss and presence of anti HBe (HBeAg seroconversion) at the end of Week 72 (48 weeks of treatment and 24 weeks of follow-up) | approximately 2.5 years
For HBeAg negative patients: Proportion of patients with HBV DNA </= 2000 IU/ml and ALT normalization | approximately 2.5 years
Safety: Incidence of adverse events | approximately 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Poland (8):
  - Bytom
  - Dębica
  - Gdansk
  - Krakow
  - Mysłowice
  - Racibórz
  - Wroclaw
  - Łańcut